CLINICAL TRIAL: NCT01714947
Title: Mass Balance, Pharmacokinetics, and Metabolism of [^14C]-Alisertib in Patients With Advanced Solid Tumors or Lymphomas
Brief Title: Mass Balance, Pharmacokinetics and Metabolism Study of Alisertib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C14014; U1111-1187-6760 (Other: WHO)
Record Dates: First submitted 2012-10-17; First posted 2012-10-26 (Estimated); Results first posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-02

CONDITIONS: Advanced Solid Tumors; Lymphoma
Keywords: Drug Therapy
MeSH Terms: conditions — Lymphoma | interventions — MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alisertib (Experimental): Part A: [^14C]-alisertib 35 mg, oral solution containing 80 - 100 microcuries (μCi) of total radioactivity (1.19 - 1.48 mCi/mmol), orally, single dose on Day 1.
  Part B: Alisertib 50 mg, enteric coated tablets, orally, twice daily for 7 days, followed by 14-day washout period in 21-day cycles until disease progression or unacceptable treatment-related toxicity (Up to 3 Cycles).
  Interventions: Drug: [^14C]-alisertib; Drug: alisertib

INTERVENTIONS:
Drug: [^14C]-alisertib — [^14C]-alisertib oral solution
  Other Names: MLN8237
Drug: alisertib — Alisertib enteric coated tablets
  Other Names: MLN8237

SUMMARY:
The purpose of this study is to assess the mass balance (i.e. cumulative excretion of total radioactivity [TRA] in urine and feces) of alisertib and pharmacokinetic (PK) of alisertib in plasma and urine, and of TRA in plasma and whole blood.

DETAILED DESCRIPTION:
The drug being tested in this study is called alisertib (MLN8237). Alisertib is being tested to treat participants who have advanced solid tumors or lymphomas. This study looked at mass balance, pharmacokinetics (PK), metabolism, elimination and safety of alisertib.

The study enrolled 3 patients. The study consisted of 2 parts: Part A and Part B. Participants received:

* [^14C]-alisertib 35 mg in Part A
* alisertib 50 mg in Part B

Participants were asked to take a single dose of [^14C]-alisertib oral solution containing 80-100 μCi of total radioactivity (1.19-1.48 mCi/mmol) in Part A and alisertib 50 mg, orally, twice daily for 7 days in 21-day cycles until disease progression or unacceptable toxicity in Part B.

This single center trial was conducted in United States. The overall time to participate in this study was up to 117 days. Participants remained confined to clinic in Part A and made multiple visits to the clinic in Part B. Participants were contacted 30 days after last dose of alisertib in Part A (if not continuing in Part B), or were contacted by telephone or a final visit 30 days after receiving their last dose of alisertib in Part B for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

Each participants must meet all of the following inclusion criteria to be enrolled in the study:

* 18 years or older.
* Histologically or cytologically confirmed metastatic and/or advanced solid tumors or lymphomas for which standard curative or life-prolonging treatment does not exist, or is no longer effective or tolerable.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Expected survival longer than 3 months from enrollment in the study.
* Radiographically or clinically evaluable tumor.
* Suitable venous access for the conduct of blood sampling.
* Recovered from the reversible effects of prior antineoplastic treatment (with the exception of alopecia and Grade 1 neuropathy).
* Female participants who are postmenopausal for at least 1 year OR are surgically sterile OR if of childbearing potential, agree to practice 2 effective methods of contraception at the same time.
* Male participants who agree to practice effective barrier contraception during the entire study and through 4 months after the last dose of study drug OR agree to abstain from heterosexual intercourse.

Exclusion Criteria:

Participants meeting any of the following exclusion criteria are not to be enrolled in the study:

* Female participants who are lactating or have a positive serum pregnancy test.
* Treatment with any investigational products or systemic antineoplastic treatment within 21 days before the first dose of alisertib.
* Medical conditions requiring daily, chronic, or regular use of proton pump inhibitors(PPIs) within 7 days preceding the first dose of alisertib, or H2-receptor antagonists within 24 hours preceding the first dose of alisertib.
* Participants requiring systemic anticoagulation (excluding low-dose aspirin, or low-dose anticoagulation to maintain patency of venous access devices). Low molecular weight heparin, administered as preventive treatment, is allowed if the participant has tolerated treatment with a stable dose and schedule without bleeding complications for more than 1 month.
* Major surgery within the 14 days preceding the first dose of alisertib.
* Infection requiring systemic intravenous (IV) antibiotic therapy within 14 days preceding the first dose of study drug, or other severe infection.
* Life-threatening or uncontrolled medical illness unrelated to cancer.
* Ongoing nausea or vomiting that is Grade 2 or worse in intensity.
* Diarrhea that is Grade 2 or worse in intensity or use of an antimotility agent to control diarrhea to an intensity of Grade 1 or lower level.
* Known GI disease or GI procedures that could interfere with the oral absorption, excretion, or tolerance of alisertib.
* History of urinary and/or fecal incontinence.
* History of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness such as severe chronic obstructive pulmonary disease.
* Inability to swallow tablets, or inability or unwillingness to avoid taking anything by mouth except for water and prescribed medications for 2 hours before and 1 hour after the first dose of alisertib.
* Inadequate bone marrow or other organ function as specified in study protocol.
* Any cardiovascular condition specified in the study protocol.
* Known or suspected human immunodeficiency virus (HIV) positive or hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection.
* Inability to comply with study visits and procedures including required inpatient confinement (approximately 11-17 days).

Please note that there are additional exclusion criteria. The study center will determine if you meet all of the criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-01-24 (Actual); Primary Completion 2013-04-04 (Actual); Study Completion 2013-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Comprehensive Clinical Development, Tacoma, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 24 January 2013 to 14 June 2013.
Pre-assignment Details: Participants with a diagnosis of advanced solid tumors or lymphomas received [^14C]-alisertib 35 mg oral solution single dose in Part A and alisertib 50 mg for 7 days in 21-day cycles in Part B.
Period: Part A
Arm/Group | Alisertib
Started | 3
Completed | 3
Not Completed | 0
Period: Part B
Arm/Group | Alisertib
Started | 3
Completed | 0
Not Completed | 3
Not completed — Progressive Disease | 3

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least 1 dose of study drug.
Arm/Group | Alisertib
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (13.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic or Latino | 3
Race/Ethnicity, Customized [Number; unit: participants]
  White | 2
  Black or African American | 1
Region of Enrollment [Number; unit: participants]
  United States | 3
Height [Mean (Standard Deviation); unit: cm] | 173.5 (7.15)
Weight [Mean (Standard Deviation); unit: kg] | 80.27 (20.760)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.91 (8.346)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Alisertib and Drug-Related Material Following a Single Dose of [^14C]-Alisertib Oral Solution
Time Frame: Predose and multiple timepoints post-dose (up to 240 hours)
Population: Pharmacokinetic (PK) Population included all participants with sufficient dosing and PK concentration-time data to reliably estimate PK parameters and mass balance.
Measure: Mean (Standard Deviation); unit: nanomole (nmol)/liter (L)
Arm/Group | Alisertib
Number analyzed (Participants) | 3
nanomole (nmol)/liter (L)
  Alisertib | 2183.3 (161.97)
  Drug-Related Material | 2606.7 (228.98)

2. Primary Outcome: Tmax: Time of First Occurrence of Cmax for Alisertib and Drug-Related Material in Plasma Following a Single Dose of [^14C]-Alisertib Oral Solution
Time Frame: Predose and multiple timepoints post-dose (up to 240 hours)
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | Alisertib
Number analyzed (Participants) | 3
hr
  Alisertib | 1.00 (161.97) [0.5 to 2.0]
  Drug-Related Material | 1.00 (228.98) [0.5 to 2.0]

3. Primary Outcome: AUClast: Area Under the Concentration-Time Curve From Time 0 to Time of the Last Quantifiable Plasma Concentration for Alisertib and Drug-Related Material Following a Single Dose of [^14C]-Alisertib Oral Solution
Time Frame: Predose and multiple timepoints post-dose (up to 240 hours)
Population: PK Population included all participants with sufficient dosing and PK concentration-time data to reliably estimate PK parameters and mass balance.
Measure: Mean (Standard Deviation); unit: hour (hr)*nmol/L
Arm/Group | Alisertib
Number analyzed (Participants) | 3
hour (hr)*nmol/L
  Alisertib | 16800.0 (4936.60)
  Drug-Related Material | 37033.3 (20545.15)

4. Primary Outcome: AUC∞: Area Under the Concentration-Time Curve From Time 0 to Infinity, Calculated Using the Observed Value of the Last Quantifiable Plasma Concentration for Alisertib and Drug-Related Material Following a Single Dose of [^14C]-Alisertib Oral Solution
Time Frame: Predose and multiple timepoints post-dose (up to 240 hours)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*nmol/L
Arm/Group | Alisertib
Number analyzed (Participants) | 3
hr*nmol/L
  Alisertib | 17266.7 (5138.42)
  Drug-Related Material | 42233.3 (23302.43)

5. Primary Outcome: T1/2: Terminal Half Life for Alisertib and Drug-Related Material in Plasma Following a Single Dose of [^14C]-Alisertib Oral Solution
Time Frame: Predose and multiple timepoints post-dose (up to 240 hours)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Alisertib
Number analyzed (Participants) | 3
hour
  Alisertib | 23.40 (7.041)
  Drug-Related Material | 42.03 (25.255)

6. Primary Outcome: CL/F: Apparent Clearance After Extravascular Administration, Calculated Using the Observed Value of the Last Quantifiable Plasma Concentration for Alisertib Following a Single Dose of [^14C]-Alisertib Oral Solution
Time Frame: Predose and multiple timepoints post-dose (up to 240 hours)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Alisertib
Number analyzed (Participants) | 3
L/hr | 4.06 (25.6)

7. Primary Outcome: Ratio of Whole Blood Total Radioactivity (TRA) Cmax to Plasma TRA Cmax
Time Frame: Predose and multiple timepoints post-dose (up to 240 hours)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib
Number analyzed (Participants) | 3
ratio | 0.6550 (0.0671)

8. Primary Outcome: Ratio of Alisertib Plasma Cmax to Drug-Related Material TRA Plasma Cmax
Time Frame: Predose and multiple timepoints post-dose (up to 240 hours)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib
Number analyzed (Participants) | 3
ratio | 0.8397 (0.0589)

9. Primary Outcome: Ratio of Whole Blood TRA AUClast to Plasma TRA AUClast
Time Frame: Predose and multiple timepoints post-dose (up to 240 hours)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib
Number analyzed (Participants) | 3
ratio | 0.5950 (0.1010)

10. Primary Outcome: Ratio of Alisertib Plasma AUClast to Drug-Related Material TRA Plasma AUClast
Time Frame: Predose and multiple timepoints post-dose (up to 240 hours)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib
Number analyzed (Participants) | 3
ratio | 0.4997 (0.1364)

11. Primary Outcome: Ratio of Whole Blood TRA AUC∞ to Plasma TRA AUC∞
Time Frame: Predose and multiple timepoints post-dose (up to 240 hours)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib
Number analyzed (Participants) | 3
ratio | 0.6750 (0.0170)

12. Primary Outcome: Ratio of Alisertib Plasma AUC∞ to Drug-Related Material TRA Plasma AUC∞
Time Frame: Predose and multiple timepoints post-dose (up to 240 hours)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib
Number analyzed (Participants) | 3
ratio | 0.4490 (0.1204)

13. Primary Outcome: Fe: Fraction of Administered Dose of [^14C]-Alisertib Excreted in Urine
Time Frame: Predose and multiple timepoints post-dose (up to 240 hours)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent of dose
Arm/Group | Alisertib
Number analyzed (Participants) | 3
percent of dose | 2.650 (1.7935)

14. Primary Outcome: Fe: Fraction of Administered Dose of [^14C]-Alisertib Excreted in Feces
Time Frame: Predose and multiple timepoints post-dose (up to 240 hours)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent of dose
Arm/Group | Alisertib
Number analyzed (Participants) | 3
percent of dose | 87.833 (2.2898)

15. Primary Outcome: Ae: Amount of [^14C]-Alisertib Excreted in Urine
Time Frame: Predose and multiple timepoints post-dose (up to 240 hours)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nanogram equivalent [ng(eq)]
Arm/Group | Alisertib
Number analyzed (Participants) | 3
nanogram equivalent [ng(eq)] | 939420.7 (632770.92)

16. Primary Outcome: Ae: Amount of [^14C]-Alisertib Excreted in Feces
Time Frame: Predose and multiple timepoints post-dose (up to 240 hours)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng(eq)
Arm/Group | Alisertib
Number analyzed (Participants) | 3
ng(eq) | 31156703.0 (764243.97)

17. Primary Outcome: Percent of Total Radioactivity (TRA) in Urine and Feces
Time Frame: Predose and multiple timepoints post-dose (up to 240 hours)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent of TRA
Arm/Group | Alisertib
Number analyzed (Participants) | 3
percent of TRA | 90.500 (1.3115)

18. Primary Outcome: Fe: Fraction of Administered Dose of Alisertib Excreted in Urine
Time Frame: Predose and multiple timepoints post-dose (up to 240 hours)
Population: Participant from the PK Population, all participants with sufficient dosing and PK concentration-time data to reliably estimate PK parameters and mass balance, with data available for Fe.
Measure: Mean (Standard Deviation); unit: percent of dose
Arm/Group | Alisertib
Number analyzed (Participants) | 2
percent of dose | 0.009045 (0.000714)

19. Primary Outcome: Ae: Amount of Alisertib Excretion in Urine
Time Frame: Predose and multiple timepoints post-dose (up to 240 hours)
Population: Participants from the PK Population, all participants with sufficient dosing and PK concentration-time data to reliably estimate PK parameters and mass balance, with data available for Ae.
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Alisertib
Number analyzed (Participants) | 2
ng | 3215.0 (219.20)

20. Primary Outcome: Renal Clearance (CLR) of Alisertib
Time Frame: Predose and multiple timepoints post-dose (up to 240 hours)
Population: Participants from the PK Population, all participants with sufficient dosing and PK concentration-time data to reliably estimate PK parameters and mass balance, with data for CLR.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Alisertib
Number analyzed (Participants) | 2
L/hr | 0.000687 (0.000013)

21. Secondary Outcome: Percentage of Alisertib Metabolites in Plasma Following a Single Dose of [^14C]-Alisertib Oral Solution
Description: Total radioactive peak distributions of metabolites in 0 to 192 hours pooled plasma samples from participants.
Time Frame: Predose and multiple timepoints post-dose (0 to 192 hours)
Population: as for outcome 3
Measure: Number; unit: percent of plasma AUC0-192hr
Arm/Group | Alisertib
Number analyzed (Participants) | 3
percent of plasma AUC0-192hr
  Metabolite M1 | 12.0
  Metabolite M2 | 34.6
  Metabolite M3 | 5.6

22. Secondary Outcome: Percentage of Alisertib Metabolites in Urine Following a Single Dose of [^14C]-Alisertib Oral Solution
Description: Total radioactive peak distributions of metabolites in 0 to 192 hours pooled urine samples from participants.
Time Frame: Predose and multiple timepoints post-dose (0 to 192 hours)
Population: as for outcome 3
Measure: Number; unit: percent of dose
Arm/Group | Alisertib
Number analyzed (Participants) | 3
percent of dose
  Unknown | 0.24
  M8a | 0.28
  M9 | 0.66
  M536 | 0.14
  M1 | 0.84
  M8 | 0.37
  Others | 0.05

23. Secondary Outcome: Percentage of Alisertib Metabolites in Feces Following a Single Dose of [^14C]-Alisertib Oral Solution
Description: Total radioactive peak distributions of metabolites in 0 to 192 hours pooled fecal samples from participants.
Time Frame: Predose and multiple timepoints post-dose (0 to 192 hours)
Population: as for outcome 3
Measure: Number; unit: percent of dose
Arm/Group | Alisertib
Number analyzed (Participants) | 3
percent of dose
  M536 | 4.45
  M520a | 1.19
  M3a | 2.22
  M550 | 2.96
  M537 | 9.17
  M520b | 1.72
  M3 | 20.82
  M520c | 5.94
  Alisertib | 26.27
  M2 | 8.62
  Others | 0

24. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events and Serious Adverse Events
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A Serious Adverse Event (SAE) was defined as any AE at any dose that: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in a persistent or significant disability/incapacity or resulted in congenital anomaly/birth defect. A treatment-emergent adverse event is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From first dose of study drug through 30 days after the last dose of study drug (Up to 117 days)
Population: Safety Population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Alisertib
Number analyzed (Participants) | 3
Participants
  Any AE | 3
  SAE | 0

25. Secondary Outcome: Number of Participants With Clinically Significant Changes or Abnormalities in Clinical Laboratory Values Reported as AEs
Description: An abnormal laboratory was assessed to be an AE if the value lead to discontinuation or delay in treatment, dose modification, therapeutic intervention, or was considered by the investigator to be a clinically significant change from Baseline.
Time Frame: Part A: Day 1 and End of Study (EOS) Day 31 if not continuing to Part B, Part B: Days 8 and 15 of each cycle and EOS (Up to 117 days)
Population: Safety Population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Alisertib
Number analyzed (Participants) | 3
Participants
  Neutrophil Count Decreased | 1
  Neutropenia | 1
  Blood Magnesium Decreased | 1

26. Secondary Outcome: Number of Participants With Clinically Significant Changes or Abnormalities in Vital Sign Measurements
Description: Vital signs included body temperature, heart rate, and sitting blood pressure. The investigator determined if the changes were clinically significant.
Time Frame: Part A: Day 1 and EOS (Day 31 if not continuing to Part B), Part B: Day 1 of each cycle and EOS (Up to 117 days)
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Alisertib
Number analyzed (Participants) | 3
Participants | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 30 days after the last dose of study drug (Up to 117 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Alisertib
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alisertib (N=3)
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Pyrexia (General disorders) | 1
Chills (General disorders) | 1
Oedema peripheral (General disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Blood magnesium decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Headache (Nervous system disorders) | 1
Scrotal swelling (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.